CLINICAL TRIAL: NCT00778284
Title: Comparative, Randomized, Single-Dose, 2-Way Crossover Bioavailability Study of Ranbaxy and GlaxoSmithKline (Augmentin®) 400 mg Amoxicillin (as the Trihydrate)/57 mg Clavulanic Acid (as the Potassium Salt) Chewable Tablets in Healthy Adult Volunteers Following Administration of a Two Tablet Dose Under Fed Conditions
Brief Title: Bioequivalence Study of Amoxicillin 400 mg/Clavulanic Acid 57 mg Chewable Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA02873
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Amoxicillin 400mg + clovalunic acid 57.5mg chewable tablets of Ranbaxy
  Interventions: Drug: Amoxicillin 400mg + clovalunic acid 57.5mg chewable tablets
- 2 (Active Comparator): Augumentin chewable tablets of Glaxosmithkline
  Interventions: Drug: Amoxicillin 400mg + clovalunic acid 57.5mg chewable tablets

INTERVENTIONS:
Drug: Amoxicillin 400mg + clovalunic acid 57.5mg chewable tablets

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Ranbaxy and GlaxoSmithKline (Augmentin®) 400 mg amoxicillin (as the trihydrate) and 57 mg clavulnic acid (as the potassium salt) chewable tablet, following administration of 2 tablet dose under fed conditions

DETAILED DESCRIPTION:
The study was conducted as an open-label, randomized, 2-way crossover study to compare the single-dose relative bioavailability of Ranbaxy and GlaxoSmithKline (Augmentin® 40o mg) amoxicillin (as the trihydrate)/57 mg clavulanic acid (as the potassium salt) chewable tablet, following administration of 2 tablet dose under fed conditions A total of 40 Subjects, 20 males and 20 females; were enrolled in the study, and 39 subjects, 20 males and 19 females, completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female volunteers, 18-55 years of age
2. Weighing at least 52 kg for males and 45 kg for females and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983);
3. Medically healthy subjects with clinically normal laboratory profiles;
4. Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the study and throughout the study or be using one of the following acceptable birth control methods:

   surgically sterile (bilateral tubal ligation, hysterectomy bilateral oophorectomy) 6 months minimum; IUD in place for at least 3 months; barrier methods (condom, diaphragm) with spermicide for at least 14 days pror to the start of the study and .throughout the study; surgical sterilization of the partner (vasectomy for 6 months minimum); hormonal contraceptives for at least 3 months pdor to the start of the study. Other birth control methods may be deemed acceptable. Postmenopausal women with amenorrhea for at least 2 years will be eligible;
5. Voluntarily consent to participate in the study.

Exclusion Criteria:

Subject candidates must not be enrolled in the study if they meet any of the following criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic,gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
2. In addition, history or presence of:

   alcoholism or drug abuse within the past 2 years; hypersensitivity or idiosyncratic reaction to antibiotics, especially penicillins, cephalosporins and amoxicillin and/or clavulanic acid
3. Female subjects who are pregnant or lactating.
4. Subjects who have been on an abnormal diet (for whatever reason) during the 30 days prior to the first dose.
5. Subjects who have made a donation (standard donation amount or more) of blood or blood products (with the exception of plasma as noted below) within 30 days prior to the study.
6. Subjects who have made a plasma donation within 7 days prior to the study
7. Subjects who have participated in another clinical trial within 30 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-10; Primary Completion 2002-10 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html